CLINICAL TRIAL: NCT03682211
Title: Intranasal Fentanyl Versus Intravenous Morphine in the Emergency Department Treatment of Severe Painful Sickle Cell Crises in Children
Brief Title: Intranasal Fentanyl Versus Intravenous Morphine in the Treatment of Severe Painful Sickle Cell Crises in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: National Children's Research Centre (Unknown); Our Lady's Children's Hospital, Crumlin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCC01; 2011-005161-20 (EudraCT Number); ISRCTN67469672 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2018-09-11; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Pain; Sickle Cell Disease
Keywords: Sickle cell disease; Paediatric; Pain; Analgesia; Intranasal; Fentanyl
MeSH Terms: conditions — Pain; Anemia, Sickle Cell; Agnosia | interventions — Fentanyl; Morphine

STUDY DESIGN:
Intervention Model Description: randomised, double-blind, double-dummy active control trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: All clinical and research staff, patients and parents are blinded to the treatment allocation. All study drugs will be packaged in blinded trial packs by a clinical trial pharmacist who is blinded to interventions and outcomes.The matched size and shape of the placebo ampoule is necessary to maintain blinding of intervention by the investigators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Intranasal Fentanyl (Experimental): Subjects will receive 50 μg/ml intranasal fentanyl citrate and a placebo matched to intravenous morphine (1 ml water for injection) at time 0
  Interventions: Drug: Fentanyl Citrate
- Active IV Morphine (Active Comparator): Subjects will receive 10 mg/ml intravenous morphine sulphate and a placebo matched to intranasal fentanyl (2 ml water)
  Interventions: Drug: Morphine sulphate

INTERVENTIONS:
Drug: Fentanyl Citrate — 50 μg/ml fentanyl citrate (Sublimaze, Janssen Cilag, Ltd, Marketing Authorisation No. PA 0748/044/001) administered intranasally using the MAD Nasal Intranasal Mucosal Atomiser Device
  Other Names: Fentanyl; Sublimaze
  Arms: Active Intranasal Fentanyl
Drug: Morphine sulphate — 10 mg/ml Morphine sulphate BP (Antigen Pharmaceuticals, Marketing Authorisation No.PA 73/20/1) administered intravenously.
  Other Names: Morphine sulfate; Morphine
  Arms: Active IV Morphine

SUMMARY:
Sickle cell anaemia is an inherited blood disorder which results in abnormal sickle shaped red blood cells which do not fit well through small blood vessels. These blockages prevent oxygen (in blood) from reaching different parts of the body resulting in painful crisis. This study will compare the effectiveness of two types of pain medication, one given through a vein and one squirted up the nose.

DETAILED DESCRIPTION:
Children with sickle cell disease (SCD) frequently and unpredictably present to the emergency department (ED) with pain. The painful event is the hallmark acute clinical manifestation of SCD, characterised by sudden onset and is usually bony in origin. This study aims to establish if 1.5mcg/kg of intranasal fentanyl (INF; administered via a Mucosal Atomiser Device, MAD™) is non-inferior to intravenous morphine 0.1 mg/kg in severe SCD-associated pain.

This study is a randomised,double-blind, double-dummy active control trial of children (weighing more than 10 kg) between 1 year and 21 years of age with severe painful sickle cell crisis. Severe pain is defined as rated seven or greater on a 0 to 10 age-appropriate numeric pain scale or equivalent. The trial will be conducted in a single tertiary urban paediatric ED in Dublin, Ireland. Each patient will receive a single active agent and a single placebo via the intravenous and intranasal routes. All clinical and research staff, patients and parents will be blinded to the treatment allocation. The primary endpoint is severity of pain scored at 10 min from administration of the study medications. Secondary endpoints include pain severity measured at 0, 5, 15, 20, 30, 60 and 120 min after the administration of analgesia, proportion of patients requiring rescue analgesia and incidence of adverse events. The trial ends at 120 min after the administration of the study drugs. A clinically meaningful difference in validated pain scores has been defined as 13 mm. Setting the permitted threshold to 50% of this limit (6 mm) and assuming both treatments are on average equal, a sample size of 30 patients (15 per group) will provide at least 80% power to demonstrate that INF is non-inferior to IV morphine with a level of significance of 0.05.

This clinical trial will inform of the role of INF 1.5mcg/kg via MAD in the acute treatment of severe painful sickle cell crisis in children in the ED setting.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1 - 21 years
* Weight ≥10 kg and ≤70 kg
* Known sickle cell disease presenting with severe pain
* Written informed consent, ideally from both parents (and assent, where appropriate), obtained prior to painful crisis (for example, in Haematology clinic)
* Verbal consent (and assent, where appropriate) obtained at the time of the painful crisis in the ED
* Hospital admission required for painful crisis

Exclusion Criteria:

* Patient has received parenteral narcotic analgesic within 4 hours of ED presentation
* Oxygen saturations below 95% on initial assessment
* Altered conscious state as defined by a Glasgow Coma score less than 15
* Contraindications to fentanyl/morphine usage
* Inability to secure IV access
* Patient has participated in another clinical trial involving an Investigation Medicinal Product (IMP) within 4 weeks of dosing, or is currently enrolled in another clinical trial involving an IMP, or has been previously enrolled in this trial
* Patients who have any condition that would make him/her, in the opinion of the Investigator or Sponsor, unsuitable for the study, or who are, in the opinion of the Investigator, not likely to complete the study for any reason
* Blocked or traumatised nose

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2013-11-14 (Actual); Study Completion 2013-11-14 (Actual)

PRIMARY OUTCOMES:
Pain score as measured using the Faces, Legs, Activity, Cry, Consolability (FLACC) scale and Manchester Pain Ruler. | 10 minutes
  Severity of pain as measured using a validated pain score (visual analogue scale) at 10 minutes after administration of the intervention. The the Faces, Legs, Activity, Cry, Consolability (FLACC) scale and Manchester Pain Ruler will be used as age-appropriate pain scales for pre-verbal/early verbal children and older verbal children respectively.

SECONDARY OUTCOMES:
Pain score as measured using the Faces, Legs, Activity, Cry, Consolability (FLACC) scale and Manchester Pain Ruler. | 0, 5, 15, 20, 30, 60 and 120 minutes
  Severity of pain as measured using a validated pain score (visual analogue scale) at 0, 5, 15, 20, 30, 60 and 120 minutes after administration of the intervention. The the Faces, Legs, Activity, Cry, Consolability (FLACC) scale and Manchester Pain Ruler will be used as age-appropriate pain scales for pre-verbal/early verbal children and older verbal children respectively.
The proportion of participants requiring rescue opioid requirement. | 120 minutes
  The proportion of patients requiring rescue opioid analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Our Lady's Children's Hospital, Crumlin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barrett MJ, Cronin J, Murphy A, McCoy S, Hayden J, an Fhaili S, Grant T, Wakai A, McMahon C, Walsh S, O'Sullivan R. Intranasal fentanyl versus intravenous morphine in the emergency department treatment of severe painful sickle cell crises in children: study protocol for a randomised controlled trial. Trials. 2012 May 30;13:74. doi: 10.1186/1745-6215-13-74. PMID 22647439